CLINICAL TRIAL: NCT06924606
Title: A Phase II Study of JS207 (PD-1/VEGF Dual Antibody) in Combination With or Without JS004 or Docetaxel in Advanced Non-small Cell Lung Cancer With Disease Progression During or After the Treatment of Platinum-based Chemotherapy and Immunotherapy
Brief Title: Evaluating the Preliminary Efficacy and Safety of JS207 in NSCLC After Progression Following Platinum-based Chemotherapy and Immunotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS207-004-II-NSCLC
Record Dates: First submitted 2025-04-06; First posted 2025-04-11 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Advanced NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Patients receive JS207 10mg/kg or other dosage and docetaxel 75mg/m2, q3w.
  Interventions: Drug: JS207 injection +docetaxel
- Arm B (Experimental): Patients receive JS207 10mg/kg or other dosage and JS004 200mg, q3w.
  Interventions: Drug: JS207 injection +JS004 injection
- Arm C (Experimental): Patients receive JS207 10mg/kg or other dosage .
  Interventions: Drug: JS207 injection

INTERVENTIONS:
Drug: JS207 injection +docetaxel — Patients receive JS207 10mg/kg or other dosage and docetaxel 75mg/m2, q3w.
  Arms: Arm A
Drug: JS207 injection +JS004 injection — Patients receive JS207 10mg/kg or other dosage and JS004 200mg, q3w.
  Arms: Arm B
Drug: JS207 injection — Patients receive JS207 10mg/kg or other dosage.
  Arms: Arm C

SUMMARY:
This is a multiple-arm, open phase II clinical trial evaluating the safety, tolerability,and preliminary efficacy of JS207 in NSCLC after progression following Platinum-based chemotherapy and immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed locally advanced (stage IIIB/IIIC) NSCLC that is not amenable to radical surgery or radical radiochemotherapy, or Metastatic or recurrent NSCLC.
2. Subjects with unresectable locally advanced or metastatic or recurrent NSCLC who have failed first-line treatment with PD-1/PD-L1 inhibitors combined with platinum-based doublet chemotherapy (excluding docetaxel); or who have failed sequential first- and second-line treatment with PD-1/PD-L1 inhibitors followed by platinum-based doublet chemotherapy (excluding docetaxel).
3. Subjects must have at least one measurable lesion according to RECIST v1.1.

Exclusion Criteria:

1. Histopathologically or cytopathologically confirmed to have combined neuroendocrine component.
2. Sensitivity mutation of EGFR or ALK fusion.
3. Tumor encircles important blood vessels or has obvious necrosis and air space, and the investigator considers that it may cause hemorrhage risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-06-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1.5years
  According to the efficacy evaluation criteria for solid tumors version 1.1 (RECIST V1.1): to evaluate objective response rate (ORR)

SECONDARY OUTCOMES:
Disease control rate (DCR) | 2years
  According to the efficacy evaluation criteria for solid tumors version 1.1 (RECIST V1.1): to evaluate disease control rate (DCR)
Duration of response (DOR) | 2years
  According to the efficacy evaluation criteria for solid tumors version 1.1 (RECIST V1.1): to evaluate duration of response (DOR)
Progression-free survival (PFS) | 1.5years
  According to the efficacy evaluation criteria for solid tumors version 1.1 (RECIST V1.1): to evaluate progression-free survival (PFS)
Overall survival (OS) | 2years
  To evaluate overall survival (OS)
AE | 2years
  Incidence and serverity of adverse events(AE),abnormal changes in laboratory and other tests with clinical significance
Abnormal changes in laboratory | 2years
  Incidence and serverity of abnormal changes in laboratory and other tests with clinical significance

OTHER OUTCOMES:
the trough concentrations (PK) | 1.5years
  to characterize the tough concentration of JS207&JS004
Neutralizing antibody(Nab) | 1.5years
  to characterize the neutralizing antibody of JS207&JS004
Antidrug antibodies (ADA) | 1.5years
  to characterize antidrug antibodies of JS207&JS004

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Jilin Cancer Hospital, Jilin, Changchun
  - Hunan Cancer Hospital, Hunan, Changsha
  - West China Hospital, Sichuan University, Sichuan, Chengdu
  - Second Affiliated Hospital, PLA Academy of Military Medical Sciences, Chongqing, Chongqing Municipality
  - Army Medical Center, PLA, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangdong, Guangzhou
  - Harbin Medical University Cancer Hospital, Heilongjiang, Harbin
  - Anyang Tumor Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - The First People's Hospital of Changde, Changde, Hunan
  - The First Affiliated Hospital of Nanchang University, Jiangxi, Nanchang
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - The Third People's Hospital of Datong, Datong, Shanxi
  - Yibin Second People's Hospital, Yibin, Sichuan
  - Affiliated Tumor Hospital of Xinjiang Medical University, Xinjiang, Xinjiang
  - Shanghai Pulmonary Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No